CLINICAL TRIAL: NCT02337348
Title: Optical Coherence Tomography (OCT) Guided Compared to Conventional Angiography Guided Coronary Intervention in Stentfailure
Brief Title: Prospective Randomized Optical Coherence Tomography Oslo tRial
Acronym: PROCTOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to slow inclusion
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Eigil Fossum, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013/1653/REK
Record Dates: First submitted 2014-12-23; First posted 2015-01-13 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Myocardial Infarction; Angina
Keywords: coronary stents
MeSH Terms: conditions — Myocardial Infarction; Angina Pectoris | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OCT guided coronary intervention (Experimental): Coronary angiography and optical coherence tomography imaging
  Interventions: Other: Optical coherence tomography; Radiation: Coronary angiography
- Conventional coronary intervention (Active Comparator): Coronary angiography
  Interventions: Radiation: Coronary angiography

INTERVENTIONS:
Other: Optical coherence tomography — Preintervention imaging
  Other Names: OCT
  Arms: OCT guided coronary intervention
Radiation: Coronary angiography — Conventional coronary intervention

SUMMARY:
Coronary artery intervention with stents is a routine procedure with several clinical indications. A stentfailure, ie stentrestenosis and/or stentthrombosis will occur in some patients. Several different mechanisms have been suggested. Stentfailure may be caused by mechanical properties of the stent. This may be secondary to suboptimal stentimplantation, ie over/undersizing or acquired ie malapposition or stentfracture. These stentproperties may be difficult to identify with conventional coronary angiography due to low image resolution. The hypothesis of the study is that high resolution imaging with optical coherence tomography (oct) will improve diagnosis and enable a more specific or tailored treatment with a subsequent reduction in later stentfailure.

DETAILED DESCRIPTION:
The hypothesis of the PROCTOR study is that high resolution imaging with optical coherence tomography (oct) will improve diagnosis and enable a more specific or tailored treatment in stent failure. However, the prevalence of stentfailure (ie stent malapposition, stentfracture, stentedgedissections etc) not causing clinical endpoints is not known. In a subset of patients (n=100) with previously implanted stents performing a new coronary angiography based on clinical indication, functional or patent stents (decided by Heart team) will be characterized with OCT and the patients followed for 5 years. The purpose of this substudy, OCT IPS (OCT In Patent Stents), is to estimate the prevalence of stentpathology in patent or functional stents and compare findings with the active arm of PROCTOR.

ELIGIBILITY:
Inclusion Criteria:

Clinical indication for coronary angiography and intervention due to stentfailure, both stentrestenosis and stentthrombosis in stable patients or unstable patients with acute coronary syndrome.

Exclusion Criteria:

* Patient not able to give informed consent.
* Unwillingness.
* Life expectancy < 5 years.
* Reduced kidney function with GRF<45.
* Coronary artery diameter < 2.5mm.
* Pregnancy.
* Patients without 11-digit Norwegian personal number.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2014-08; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Target lesion revascularisation | 5 years

SECONDARY OUTCOMES:
non-fatal myocardial infarction | 5 years
Cardiovascular mortality | 5 years

OTHER OUTCOMES:
Change in kidney function | 5 years
  Number of participants with more than 25% increase in serum creatinin.

CONTACTS AND LOCATIONS:
Overall Officials: Eigil Fossum, MD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo university hospital, Oslo, Norway